CLINICAL TRIAL: NCT00434525
Title: Metabolic Effects of Laparoscopic Sleeve Gastrectomy With or Without Omentectomy: Prospective Randomized Trial
Brief Title: Laparoscopic Sleeve Gastrectomy With and Without Omentectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Esteban Varela MD, MPH, VA North Texas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-011
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-08

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Bariatric Surgery; Obesity Surgery; Omentectomy; Sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Sleeve gastrectomy with omentectomy (Experimental)
  Interventions: Procedure: Laparoscopic restrictive procedure
- 2 Sleeve gastrectomy (Active Comparator)
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic restrictive procedure — Patients will receive laparoscopic sleeve gastrectomy with or without omentectomy
  Arms: 1 Sleeve gastrectomy with omentectomy
Procedure: Sleeve gastrectomy — Sleeve gastrectomy
  Arms: 2 Sleeve gastrectomy

SUMMARY:
* The investigators aim to determine the clinical and metabolic effects of sleeve gastrectomy with or without omentectomy in the treatment of morbid obesity.
* The investigators hypothesize that the endocrine suppression of ghrelin (appetite hormone)and resistin (insulin antagonist) provided by sleeve gastrectomy and omentectomy (omentum or intra-abdominal fat removal) will provide clinical and metabolic benefits for morbidly obese patients.

DETAILED DESCRIPTION:
This is a phase 3 prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese VETERANS ONLY (BMI>35 with comorbidities or BMI>40)
* Age > 18

Exclusion Criteria:

* Pregnancy
* Uncontrolled medical or psychiatric conditions
* Previous bariatric procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Weight loss | 5 years

SECONDARY OUTCOMES:
Metabolic outcomes | 5 years
Diabetes resolution | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Varela, MD, MPH, Principal Investigator — VA North Texas
Locations (1):
- VA North Texas, Dallas, Texas, United States